CLINICAL TRIAL: NCT00168155
Title: Phase 2 Study of Neoadjuvant 5-FU + Leucovorin + CPT-11 in Patients With Resectable Liver Metastases From Colorectal Adenocarcinoma
Brief Title: Study of 5-FU + Leucovorin + CPT-11 in Patients With Resectable Liver Metastases From Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Collaborators: Pfizer (Industry)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTAIV-0020-357
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Adenocarcinoma; Liver Metastases
Keywords: resectable liver metastases; colorectal adenocarcinoma; survival; neoadjuvant chemotherapy

INTERVENTIONS:
Drug: perioperative chemotherapy

SUMMARY:
When colon or rectal cancer has spread to the liver, the cancer in the liver can sometimes be removed surgically. However, the cancer has a chance or reoccurring in the liver or elsewhere in the body. This study will determine if giving chemotherapy treatment before the surgery can reduce the chances that the cancer will come back.

DETAILED DESCRIPTION:
When colon or rectal cancer has spread to the liver, the cancer in the liver can sometimes be removed surgically. However, the cancer has a chance or reoccurring in the liver or elsewhere in the body. This study will determine if giving chemotherapy treatment before the surgery can reduce the chances that the cancer will come back.

ELIGIBILITY:
Inclusion Criteria:

* stage IV colorectal cancer isolated to the liver
* one measurable lesion
* metastases are completely resectable or amenable to ablation
* Karnofsky >70
* Adequate bone marrow function
* adequate hepatic function
* adequate renal function
* informed consent

Exclusion Criteria:

* primary tumor not controlled by locoregional treatments
* bilateral portal vein and/or hepatic artery involvement
* previous chemotherapy directed at treatment of metastatic colorectal cancer
* underlying acute or chronic liver disease
* Gilbert's disease
* patients receiving phenytoin or phenobarbital prophylaxis
* presence of any concurrent medical or psychiatric condition that serves as a contraindication to surgery or chemotherapy
* pregnancy
* malignancy other than basal cell or squamous cell carcinoma of the skin within the preceding 5 years
* use of another investigational medication concurrently or within 4 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2002-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bathe, MD, Principal Investigator — Alberta Health services
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Bathe OF, Ernst S, Sutherland FR, Dixon E, Butts C, Bigam D, Holland D, Porter GA, Koppel J, Dowden S. A phase II experience with neoadjuvant irinotecan (CPT-11), 5-fluorouracil (5-FU) and leucovorin (LV) for colorectal liver metastases. BMC Cancer. 2009 May 20;9:156. doi: 10.1186/1471-2407-9-156. PMID 19457245